CLINICAL TRIAL: NCT02382965
Title: Transcranial Focused Ultrasound for Deep Brain Stimulation in Humans
Brief Title: Ultrasound in Deep Brain Stimulation
Status: Terminated | Type: Observational
Why Stopped: PI left University no data available
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1501M61441
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Sub-cortical Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ultrasound
  Interventions: Device: transcranial focused ultrasound

INTERVENTIONS:
Device: transcranial focused ultrasound

SUMMARY:
It is the purpose of this proposal to apply tFUS to the ventral posterior lateral (VPL) nucleus of the thalamus in humans.

DETAILED DESCRIPTION:
Current non-invasive neuromodulatory approaches like transcranial magnetic stimulation (TMS) and transcranial direct current stimulation (tDCS) have proven efficacious for inducing transient plastic changes in the human cortex. However, these technologies have poor spatial resolution, suffer from a depth focality tradeoff and experience significant attenuation at depth. Thus, they cannot effectively target neural tissue below the surface of the cortex. Transcranial focused ultrasound (tFUS) is a new and very promising non-surgical low-energy technique for inducing transient plasticity with high spatial resolution, adjustable focus and low tissue attenuation. tFUS has been used safely and effectively for neural stimulation in mouse, rabbit and monkey and my research has shown tFUS to also be a safe and effective method of transient cortical stimulation in humans. Having demonstrated its efficacy in humans for cortical stimulation, the next step is to take advantage of tFUS' high spatial resolution and deep focal lengths to stimulate sub-cortical neural structures. Currently, the only way to stimulate sub-cortical structures involves expensive and risky surgery. It is the purpose of this proposal to test tFUS for sub-cortical stimulation. The ability to individually stimulate small neural structures deep to the cortex without invasive surgery would have broad application in basic neuroscience for the investigation of brain structure and function as well as for the potential diagnosis and therapy of many neurological and psychiatric diseases.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age
* Provide written informed consent

Exclusion Criteria:

* Evidence of a current significant medical illness or psychiatric or central or peripheral neurologic disorder
* History of loss of consciousness of more than ten minutes in the past year or loss of consciousness in a lifetime that required rehabilitation services
* Personal or family history of seizure
* Any history of stroke/transient ischemic attack (TIA)
* Taking any medications that may decrease the threshold for seizure
* Affirmative answers to one or more questions of the provided attached safety questionnaires. These are not absolute contraindications to this study but the risk/benefit ratio will be carefully balanced by the PI
* Failure to follow laboratory or study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults will be enrolled for Transcranial Focused Ultrasound for Deep Brain Stimulation
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Somatosensory evoked potential amplitude | one year